CLINICAL TRIAL: NCT05274165
Title: Evaluation of New Fitting Characteristics for Extended Wear Hearing Aid Technology- Trial to Success Rate
Brief Title: Evaluation of New Fitting Characteristics for Extended Wear Hearing Aid Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Sound Relief Tinnitus & Hearing Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-504
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: In this study, new hearing aid candidates will be randomly assigned to one of two groups, but such that each group will have an equal number of participants.
Who Masked: Participant
Masking Description: Participants will not know which device they are wearing as these devices are placed deep in the ear canal by a licensed hearing care professional. The devices are designed to stay in the ear 24 hours a day, and can be worn for several weeks or months at a time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Participants will be fit with commercially available Lyric devices, which range from size XXS to XXL.
  Interventions: Device: Lyric Hearing Aid- Commercially Available
- Group B (Experimental): Participants will be fit either with the commercially available Lyric devices OR devices which are designed with a new fitting characteristic. This increases the pool of sizes from which the hearing care professional can choose to fit participant.
  Interventions: Device: Lyric Hearing Aid- Experimental Design; Device: Lyric Hearing Aid- Commercially Available

INTERVENTIONS:
Device: Lyric Hearing Aid- Experimental Design — Extended wear hearing aid with a fitting modification that is currently not available
  Arms: Group B
Device: Lyric Hearing Aid- Commercially Available — Extended wear hearing aid that is currently available

SUMMARY:
Two groups of hearing aid candidates will be fit with extended wear technology. One group will be fit with the commercially available models, and the other group will be fit with either the commercially available model or a new model with different fitting characteristic.

After an appropriate trial period, the success rate of each group will be determined by the desire to purchase devices.

DETAILED DESCRIPTION:
Hearing aid candidates will be assigned to either Group A or Group B. Group A will be fit only with extended wear devices that are commercially available. Group B will be fit with either the commercially available devices, or a set of devices that have a new fitting characteristic, depending on what is most appropriate and the best fit. Because extended wear devices are inserted by a hearing care professional and sit deep within the ear canal, participants will be blinded as to which devices they are wearing. After a typical hearing aid trial period (i.e. 30 days), participants will be asked to make a determination on whether they would purchase if given the option. The percentage of people that indicate a desire to purchase devices from Group A will be compared to the percentage of people that indicate a desire to purchase devices from Group B to determine if the offering of additional fitting options results in an increase in intent to purchase, or a trial to success rate.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hearing loss
* New hearing aid users with no previous hearing aid experience interested in trying Lyric devices
* Must meet Lyric candidacy (see exclusion criteria)

Exclusion Criteria:

* middle ear disease, including but not limited to history of tympanic membrane perforations, chronic otitis media, cholesteatoma, PE tubes
* radiation therapy to head or neck area
* participants who need regular MRI testing
* participants who regularly scuba dive or swim underwater

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sound Relief Hearing Center, Highlands Ranch, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 12 | 13
Completed | 9 | 10
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Participants who met the fitting criteria for the Lyric extended wear hearing device
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Customized [Mean (Full Range); unit: years] | 62 [51 to 77] | 66 [57 to 75] | 64 [51 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 9 | 6 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Trial to Success Rate
Description: Percentage of participants who express intent to purchase devices at end of study trial period. No statistical analysis was performed on this outcome measure.
Time Frame: Day 30 of study
Population: All participants that were fit with extended wear hearing devices
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 9 | 10
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Group A: Participants for whom only the commercially available Lyric sizes were available. The clinician was limited to choosing the best fit among the commercially available sizes only. This group includes participants who started and ended the trial with only commercially available sizes of Lyric.
- Group B: Participants for whom the commercially available sizes and the experimental sizes of Lyric were available. The clinician was able to choose the best fit from all sizes. This group includes participants who may have started the trial with an experimental device but ended with a commercially available size, and vice-versa, depending on the wearing comfort and the discretion of the clinician.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 1/12 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=12) | Group B (N=13)
discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Discomfort and redness of middle ear tissue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT05274165/Prot_SAP_000.pdf